CLINICAL TRIAL: NCT02033668
Title: A Randomized, Open Label, Parallel-Group Study to Estimate Bioavailability and to Assess the Pharmacokinetic Profile, Safety and Tolerability of GSK933776 Administered by Subcutaneous or Intramuscular Injection Relative to Intravenous Administration to Healthy Volunteers
Brief Title: Pharmacokinetic (PK) Study of GSK933776 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 116891
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Atrophy, Geographic
Keywords: bioavailability; Pharmacokinetics; intravenous; subcutaneous and intramuscular administration; amyloid beta; monoclonal antibody
MeSH Terms: conditions — Geographic Atrophy; Plaque, Amyloid | interventions — Organization and Administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A (Active Comparator): Participants in this arm will receive single 200 milligram (mg) dose of GSK933776 administered by IV infusion
  Interventions: Drug: GSK933776 for IV administration
- Arm B (Experimental): Participants in this arm will receive single 200 mg dose of GSK933776 administered SQ
  Interventions: Drug: GSK933776 for SQ administration
- Arm C (Experimental): Participants in this arm will receive 50 mg dose of GSK933776 administered SQ once weekly for 4 weeks (total dose = 200 mg).
  Interventions: Drug: GSK933776 for SQ administration
- Arm D (Experimental): Participants in this arm will receive single 200 mg dose of GSK933776 administered IM
  Interventions: Drug: GSK933776 for IM administration

INTERVENTIONS:
Drug: GSK933776 for SQ administration — Antibody solution for subcutaneous injection with unit dose strength of 50mg/mL administered as 200 mg single dose or as repeat dose of 50 mg weekly for 4 weeks
  Arms: Arm B; Arm C
Drug: GSK933776 for IM administration — Antibody solution for intramuscular injection with unit dose strength of 50mg/mL administered as 200 mg single dose
  Arms: Arm D
Drug: GSK933776 for IV administration — Antibody solution for intravenous injection with unit dose strength of 50mg/mL administered as 200 mg single dose through an IV catheter over approximately 1 hour
  Arms: Arm A

SUMMARY:
This study is intended to enable a possible transition to intramuscular (IM) or subcutaneous (SQ) administration for subsequent studies with GSK933776 by characterizing the safety, tolerability, PK and pharmacodynamic profiles, and immunogenicity of GSK933776 following IM and SQ administration in healthy volunteers. Such alternate routes of administration may provide more options in the selection of an efficacious dose for subsequent development in patients with geographic atrophy. There will be four treatment arms in the study and participants will be assigned to 1 of 4 possible treatment arms in a 1:1:1:1 ratio. The planned number of evaluable participants for this study is 24 with 6 participants completing all critical assessments in each of the four treatment arms. The total duration of participation from screening to follow-up for Treatment Arms A, B and D (single dose of GSK933776), will be approximately 113 days and total duration for Treatment Arm C (repeat dose of GSK933776) will be approximately 134 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject 18 to 50 years of age at the time of signing the informed consent
* In general good health as determined by a physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the condition is unlikely to introduce additional risk factors and will not interfere with the study procedures
* Body weight >=55 kilograms (kg) (121 pounds [lbs]) and <=85 kg (187 lbs) with a body mass index (BMI) between 18.5 and 29 kg per meter square (inclusively) at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 milli international unit (MIU)/milliliter (mL) and estradiol <40 picogram/mL (<140 picomoles/Liter) is confirmatory.
* Male subjects must agree to use one form of acceptable contraception methods if their partner is of childbearing potential. This criterion must be followed from the time of the screening visit through the follow up visit (84 days after last dose of study medication).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Known risk history of Central nervous system (CNS) disorders: History and/or evidence (computed tomography or magnetic resonance imaging scan performed within the past 12 months) of cerebral haemorrhage OR a known risk of cerebral haemorrhage, including uncontrolled hypertension, cerebrovascular malformation, coagulopathy, central nervous system (CNS) vasculitis, degenerative or inflammatory/demyelinating CNS conditions or any other condition that the Investigator and/or the medical monitor considers as a relevant risk factor for cerebral haemorrhage. Transient ischemic attack (TIA)/cerebrovascular accident (CVA) in the last year, or other uncontrolled risk factors for stroke; History of seizures (except febrile seizures in childhood) or recent unprovoked seizure; Uncontrolled type 2 diabetes mellitus (glycated hemoglobin >10%), active cardiovascular disease (e.g., moderate-severe angina, unstable angina, myocardial infarction (MI) within the last 2 years, symptomatic congestive heart failure, clinically significant arrhythmia); Current blood clotting or bleeding disorder or conditions that predispose to these (e.g. cancer); Diagnosis of currently active, or, in remission but chronic relapsing, systemic autoimmune disease or condition (e.g. multiple sclerosis, lupus erythematosus etc) that the Investigator and/or the medical monitor considers as a relevant risk factor for concomitant administration of a therapeutic monoclonal antibody.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Use of prescription drugs or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* A positive pre-study drug/alcohol screen. Current or recent drug or alcohol abuse or dependence. History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 units for males or >7 units for females. One drink is equivalent to 12 gram (g) of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits. Use of illegal drugs.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates their participation.
* Seated systolic blood pressure >140 millimeter of mercury (mmHg) or seated diastolic blood pressure of > 90 mmHg
* QTc >450 millisecond (msec).
* Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) >= 2xupper limit of normal (ULN); alkaline phosphatase and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Significant abnormalities on hematology screen: clinically significant anemia (i.e. hemoglobin <11 g/deciliter [dL] for males or <10 g/dL for females), or platelet counts below 124 Giga/L; International Normalized Ratio > 2.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive test for human immunodeficiency virus antibody
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Exposure to more than four new chemical entities within 12 months prior to screening.
* Prior allergic reactions to biological products (vaccines, antibodies) or known hypersensitivity to any of the components of the drug formulation.
* Prior participation in clinical investigations involving therapeutic monoclonal antibodies with a similar mode of action or proteins derived from monoclonal antibodies with any risk of cross- reactivity or any investigations of treatments or use of any other investigational medication or device within 2 months prior to screening or within 5 half-lives of use of such a medication prior to screening, whichever is longer.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-01-22 (Actual); Primary Completion 2014-07-15 (Actual); Study Completion 2014-07-15 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability of GSK933776 after single dose SQ or IM administration as compared to IV infusion | Blood samples will be collected at following time points: pre-dose and at (0.25, 0.5, 0.75, 1, 2, 4 hours only for IV infusion), 6, 24, 48, 72, 96, 120, 216, 336, 504, 672, 1344 and 2016 hours post dose
  Bioavailability is defined as the rate and extent to which drug reaches the systemic circulation. The relative bioavailability will be calculated from the ratio of area under concentration time curve from time zero to infinity (AUC [0-infinity]) following single dose SQ and IM injection to intravenous (IV) infusion
Relative bioavailability of GSK933776 after repeat dose SQ administration as compared to IV infusion | Blood samples will be collected at following time points: pre-dose, 6, 24, 48, 72, 96 and 120 hours post dose in each of the 4 dosing weeks and additionally at 216, 336, 504, 672, 1344 and 2016 hours post last dose
  Bioavailability is defined as the rate and extent to which drug reaches the systemic circulation. The relative bioavailability will be calculated from the ratio of AUC (0-infinity) following SQ repeat dose injections to intravenous (IV) infusion

SECONDARY OUTCOMES:
Composite of PK parameters of GSK933776 following single dose IM and SQ administration as compared to IV administration | Samples will be collected at following time points: pre-dose and at (0.25, 0.5, 0.75, 1, 2, 4 hours only for IV infusion), 6, 24, 48, 72, 96, 120, 216, 336, 504, 672, 1344 and 2016 hours post dose
  PK parameters include: area under the concentration-time curve over the dosing interval (AUC[0-tau]), maximum concentration (Cmax), time of occurrence of Cmax (Tmax), terminal phase half-life (T1/2), clearance, and volume of distribution as data permit
Composite of PK parameters of GSK933776 following repeat dose SQ administration as compared to IV administration | Blood samples will be collected at following time points: pre-dose, 6, 24, 48, 72, 96 and 120 hours post dose in each of the 4 dosing weeks and additionally at 216, 336, 504, 672, 1344 and 2016 hours post last dose.
  PK parameters include: AUC(0-tau), Cmax, Tmax, T1/2, clearance, and volume of distribution as data permit
Number of participants with adverse events as a measure of safety and tolerability following single dose administration | Up to 113 days
  AEs will be collected from the start of Study Treatment and until the follow-up contact
Clinical observation following IV, SQ and IM single dose administration as a measure of safety and tolerability | Up to 134 days
  AEs will be collected from the start of Study Treatment and until the follow-up contact
Clinical observation following IV, SQ and IM repeat dose administration as a measure of safety and tolerability | Up to 113 days
  Clinical observation include: physical examination, medical history, and review of concomitant medication
Vital sign measurement following single dose administration as a measure of safety and tolerability | Up to 134 days
  Vital sign measurements will include systolic and diastolic blood pressure, pulse rate, and body temperature measurement.
Vital sign measurement following repeat dose administration as a measure of safety and tolerability | Up to 134 days
  Vital sign measurements will include systolic and diastolic blood pressure, pulse rate, and body temperature measurement.
Electrocardiogram (ECG) measurement following single dose administration to assess safety and tolerability | Up to 113 days
  12-lead ECGs will be obtained at each time point during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT interval corrected for heart rate (QTc interval).
ECG measurement following repeat dose administration to assess safety and tolerability | Up to 134 days
  12-lead ECGs will be obtained at each time point during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc interval.
Clinical laboratory parameters assessment following single dose administration as a measure of safety and tolerability | Up to 113 days
  Clinical laboratory assessment include: hematology, clinical chemistry, urinalysis and additional parameters.
Clinical laboratory parameters assessment following repeat dose administration as a measure of safety and tolerability | Up to 134 days
  Clinical laboratory assessment include: hematology, clinical chemistry, urinalysis and additional parameters.
Plasma concentrations of GSK933776, total amyloid beta (AB), total AB fragments, as well as unbound concentrations of AB, fragments containing the epitope 1-22, as data permit following single dose administrationof GSK933776 | Up to 113 days
  The relationship between plasma concentration of GSK933776 and plasma concentration of total and free amyloid beta will be explored as data permit
Plasma concentration of GSK933776, AB, total AB fragments, as well as unbound concentrations of AB, fragments containing the epitope 1-22, as data permit following repeat dose administration | Up to 134 days
  The relationship between plasma concentration of GSK933776 and plasma concentration of total and free amyloid beta will be explored as data permit
Presence of antibodies to GSK933776 in serum samples following single dose administration of GSK933776 | Up to 113 days
  To characterize the immunogenicity profile of GSK933776 following IV, IM and SQ administration. Samples will be analyzed for the presence of anti-GSK933776 antibodies by immuno-electrochemiluminescent (ECL) screening and neutralization assays.
Presence of antibodies to GSK933776 in serum samples following repeat dose administration | Up to 134 days
  To characterize the immunogenicity profile of GSK933776 following IV, IM and SQ administration. Samples will be analyzed for the presence of anti-GSK933776 antibodies by immuno-electrochemiluminescent (ECL) screening and neutralization assays.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 116891 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/116891?search=study&search_terms=116891#rs
- Available data/document: Statistical Analysis Plan: 116891 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116891 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116891 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116891 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116891 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116891 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116891 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register